CLINICAL TRIAL: NCT04508569
Title: Evaluation of the Big Decisions Teen Pregnancy Prevention Intervention in Three South Texas School Districts
Brief Title: Evaluation of Big Decisions in Three South Texas School Districts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Collaborators: Healthy Futures of Texas (Unknown); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Big Decisions
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Big Decisions (Experimental)
  Interventions: Behavioral: Big Decisions
- Youth Voices (Active Comparator)
  Interventions: Behavioral: Big Decisions

INTERVENTIONS:
Behavioral: Big Decisions — Big Decisions is a promising teen pregnancy prevention intervention that consists primarily of abstinence-plus sexual health education curriculum. The intended dosage for students is 10 classroom-based sexual health lessons.

SUMMARY:
An evaluation of a promising Teen Pregnancy Prevention Curriculum, Big Decisions, in ninth grade students in three high schools in South Texas.

DETAILED DESCRIPTION:
Intervention Description Big Decisions is a promising teen pregnancy prevention intervention that consists primarily of abstinence-plus sexual health education curriculum. The intended dosage for students is 10 classroom-based sexual health lessons.

Classroom teachers, who receive three days of training on the curriculum as well as ongoing technical assistance, deliver Big Decisions lessons to 9th grade students. The lessons take place during normally scheduled classes over the course of three to five weeks. Classes include health, biology, and English. The curriculum focuses on helping youth make good decisions about their sexual health. There are three key messages: (1) having sex with someone is a big decision, (2) abstinence is the most effective way to avoid both pregnancy and sexually transmitted infections, and (3) teens who have sex need to use latex condoms correctly every time to reduce the risk of HIV and sexually transmitted infections and use contraception to prevent pregnancy.

In addition to a classroom curriculum, Big Decisions also includes a parent component offered to all families. This includes two parent workshops, a parent workbook, and homework for parents and children. The parent workshop meets twice during the period of time when students receive the classroom curriculum. The workshops last for 90 minutes, are offered in both English and Spanish, and are facilitated by district coordinators and grantee staff.

Comparison Condition Youth Voices Comparison Condition Description Youth Voices is a benign comparison intervention that meets for two class sessions over three to five weeks. Classroom teachers deliver Youth Voices to 9th grade students. Teachers deliver sessions during regularly scheduled classes similar to Big Decisions. Students in Youth Voices participate in facilitated discussions about two of seven potential discussion topics (nutrition, physical fitness and exercise, tobacco and e-cigarettes, participation in sports, driver safety, environmental health, and safety at work). Students take a vote, and they discuss the two topics with the most votes during the sessions. Classroom teachers facilitate Youth Voices. Teachers are trained to deliver both Youth Voices and Big Decisions and can deliver both programs to different classes during the same implementation period.

Behavioral Outcomes Sexual initiation, condom use at last sex, birth control use at last sex, ever pregnant or gotten someone pregnant, sex in the past three months, sex without a condom in the past three months, sex without birth control in the past three months Non-behavioral Outcomes Intentions to have sex, intentions to use a condom, intentions to use birth control Sample and Setting HealthyFutures of Texas staff recruited four high schools from three rural and semi-rural school districts in Texas for participation in the study. The program targets 9th-grade students in each district for participation. Each high school identified one course required for 9th grade students for program delivery (for example, health, biology, English). To be eligible for participation, students must (1) be in 9th grade, (2) be enrolled in one of the courses identified for program delivery, (3) have parental consent, and (4) provide student assent. The evaluation expects to enroll 2,596 students from 178 classrooms.

Research Design and Data Collection This evaluation is a cluster randomized controlled trial. Classrooms are the unit of randomization. Two of the three school districts are implementing the program and evaluation once a year and the third school district, with two high schools, is implementing each quarter of the academic year. At the beginning of each round of implementation, parents provide consent for participation. Two weeks before implementation, students provide assent and take the baseline survey. The evaluator randomizes the participating classes the week before implementation.

Youth will be surveyed at baseline, immediately post-intervention, and at 12-month follow-up. Baseline and immediate post-test surveys will be given in the classroom. Surveys will be collected using a survey link or using paper versions of the survey. The 12-month follow-up survey will take place in small group settings at the school. Absent students will be surveyed in-person individually by the district coordinator, by phone, or over the web. Teachers, district coordinators, and research staff will collect data.

Data for an implementation study designed to assess fidelity, attendance, and quality will be collected through fidelity logs, observations, and attendance sheets.

ELIGIBILITY:
Inclusion Criteria:

* Must be in ninth grade and enrolled in a participating class at a participating high school

Exclusion Criteria:

* Lack of consent or assent

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3170 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Use of condom or effective method of birth control last time you had sex | One year
  Did you use a condom or effective method of birth control the last time you had sex?

SECONDARY OUTCOMES:
intention to use condom or birth control | immediate post-test
  Do you intend to use a condom or effective method of birth control if you have sex
Frequency of communication with parents about abstinence and sex | immediate post-test
  How often do you talk to your parent or guardian about abstinence or sex

CONTACTS AND LOCATIONS:
Locations (1):
- Philliber Research and Evaluation, Accord, New York, United States

IPD SHARING:
Plan to Share IPD: No